CLINICAL TRIAL: NCT01258010
Title: Impact of Tranexamic Acid on Red Blood Cell Transfusion in Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JFH2011-001
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Neurosurgery; Orthopedic Surgery; Red Blood Cell Transfusion
Keywords: Red blood cell transfusion; Neurosurgery; Orthopedic surgery; Tranexamic acid; Surgical blood loss
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic acid (Experimental): Study subjects will be randomized to receive a bolus dose of 30 mg/kg of tranexamic acid administered over 30 minutes starting after the induction of anesthesia followed by a continuous intravenous infusion of tranexamic acid of 16 mg/kg/h administered up to 6 hours after surgery.
  Interventions: Drug: Tranexamic Acid
- Normal saline (NaCl 0.9%) (Placebo Comparator): Study subjects will be randomized to receive a bolus dose of normal saline (NaCl 0.9%) of equivalent volume administered over 30 minutes starting after the induction of anesthesia followed by a continuous intravenous infusion of NaCl 0.9% administered up to 6 hours after surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Bolus dose of 30 mg/kg of tranexamic acid followed by a continuous intravenous infusion of 16 mg/kg/h of tranexamic acid administered up to 6 hours after surgery.
  Arms: Tranexamic acid
Drug: Placebo — Bolus dose of normal saline (NaCl 0.9%) of equivalent volume followed by a continuous intravenous infusion of NaCl 0.9% administered up to 6 hours after surgery.
  Arms: Normal saline (NaCl 0.9%)

SUMMARY:
Spinal surgery may be associated with substantial blood loss which often requires erythrocyte transfusion. Transfusion of red blood cells (RBC) is not free of adverse events and has been associated with increased risks of infection, and globally higher morbidity and mortality.

Different techniques have been used to reduce perioperative blood losses and related transfusions. Tranexamic acid has been used successfully in cardiac and hepatic surgery. However, only a few studies have reported on the use of antifibrinolytic drugs in spinal surgery.

This study was designed to assess the efficacy and safety of tranexamic acid in spinal surgery for the reduction of RBC transfusion.

Hypothesis: the infusion of tranexamic acid during spinal surgery will reduce the risk of receiving a RBC transfusion and, in those patients transfused, reduce the number of blood products administered.

DETAILED DESCRIPTION:
Administration of study drug

The administration of tranexamic acid/placebo will start following the induction of general anesthesia. A bolus dose will be given intravenously over 30 minutes followed by a continuous infusion administered up to 6 hours postoperatively.

Drugs used for anesthesia and postoperative analgesia will be left to the discretion of the attending anesthesiologist. The administration of fluids (crystalloids, colloids and blood products) will be recorded.

Transfusion: The transfusion trigger will be < 80 g/L during surgery if the situation is stable. Transfusion may be initiated according to the attending anesthesiologist if the situation is unstable. In the case of massive bleeding, transfusion will follow our standard institutional protocol. The presence of microvascular bleeding at the surgical site will be assessed by the surgeon. The Cellsaver will not be used.

The transfusion trigger during the postoperative period will be < 80 g/L. Blood losses and the need for transfusion will be recorded from the moment of surgery up to 72 hours postoperatively.

Laboratory testing

Before surgery: hemoglobin and coagulogram values will be recorded.

During surgery: the patient's coagulation status will be assessed using a thromboelastograph (TEG). Thromboelastography is a simple coagulation test that enables evaluation of all components of hemostasis. TEG testing will be performed at the induction of anesthesia and every 2 hours throughout surgery. An additional blood sample for TEG analysis will be collected at the end of surgery if the previous test was performed more than an hour before the end of surgery.

After surgery: laboratory testing for hemoglobin, coagulogram, fibrinogen and d-dimer will be performed in the recovery room. Hemoglobin will also be measured on postoperative days 1, 2 and 3. Blood samples to assess cardiac troponin levels will be collected on postoperative days 1 and 2.

Ultrasound : Patients will have an ultrasound examination of the inferior limbs before discharge from the hospital to detect deep vein thrombosis.

Follow-up The presence of adverse events during the course of the hospital stay will be noted.

At 30 days, patients will be contacted by phone to detect any other adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 85 years
* Patients undergoing spinal surgery with expected significant blood loss
* American Society of Anesthesiologists physical status(ASA) I to III inclusive

Exclusion Criteria:

* Allergy to tranexamic acid
* Epilepsy
* Minimally invasive surgery
* Unwillingness to receive blood transfusion
* Known coagulopathy/hepatic disease
* Previous thromboembolic events
* Pregnancy
* Renal impairment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients transfusions | From surgery until 72 hours postoperatively
Number of red blood cell transfusions | From surgery until 72 hours postoperatively

SECONDARY OUTCOMES:
Measured blood losses | From surgery until 72 hours postoperatively
Morbidity | From surgery until 30 days postoperatively
  Deep vein thrombosis, pulmonary embolism, seizures, myocardial infarction, renal failure
Mortality | From surgery until 30 days postoperatively
Length of stay in the hospital | At time of discharge
Calculated blood losses | From surgery until 72 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Hardy, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal-Hôpital Notre-Dame, Montreal, Quebec, Canada